CLINICAL TRIAL: NCT07377708
Title: A Comparison of Autologous Platelet-Rich Plasma Dressing Versus Saline Dressing in the Management of Pediatric Heel Pad Injuries Due to Motorcycle Wheel-Spoke Trauma
Brief Title: Platelet-Rich Plasma Versus Saline Dressings in Pediatric Heel Pad Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Fatima Numeri, Professor and Head of Pediatric Surgery Department, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2023/1091/SIMS
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Wheel Spoke Injury; Heel Pad Injuries; Wound Healing
Keywords: Platelet Rich Plasma (PRP); Saline Dressing; Wound Care Trauma - Pediatric; Motorcycle Injuries; Soft Tissue Repair; Pediatric Surgery
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial, 1:1 allocation by lottery method (PRP dressing vs normal saline dressing).
Masking Description: No Blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Platelet-Rich Plasma Dressings (Experimental): Approximately 10 mL of venous blood is processed to prepare PRP, which is applied as a wound dressing for 3 days. Applied for about 4 weeks, with follow-up until 12 weeks.
  Interventions: Biological: Autologous Platelet-Rich Plasma (PRP) Dressing
- Normal Saline Dressing (Active Comparator): Conventional sterile saline dressings are applied daily over ~4 weeks, with follow-up until 12 weeks.
  Interventions: Other: Normal Saline Dressings

INTERVENTIONS:
Biological: Autologous Platelet-Rich Plasma (PRP) Dressing — Approximately 10 mL of venous blood is processed in the pathology department to prepare PRP, which is applied as a wound dressing. Dressings are applied over ~4 weeks, with outpatient follow-up until 12 weeks.
  Arms: Autologous Platelet-Rich Plasma Dressings
Other: Normal Saline Dressings — Conventional sterile normal saline dressings are applied over ~4 weeks, with outpatient follow-up until 12 weeks.
  Arms: Normal Saline Dressing

SUMMARY:
This study is testing whether autologous platelet rich plasma (PRP) dressings are more effective than normal saline dressings in treating heel pad injuries caused by motorcycle wheel spokes among children in Pakistan. PRP is prepared from a child's own blood and contains natural growth factors that may help wounds to heal faster. The study compares healing rates, reduction in wound size, and time to complete wound healing between the platelet-rich plasma and saline dressing groups.

DETAILED DESCRIPTION:
Motorcycle wheel-spoke injuries occur when the heel or foot becomes entrapped in the spokes of a moving motorcycle, frequently resulting in severe soft tissue damage in children. Healing of these injuries is often prolonged and challenging. Platelet-rich plasma (PRP), prepared from a patient's own blood, contains a high concentration of growth factors that promote tissue regeneration, angiogenesis, and wound contraction. Previous studies in adults with diabetic and chronic ulcers have demonstrated that PRP may accelerate wound healing compared with conventional dressings.

However, evidence supporting the use of PRP in the pediatric population, particularly for heel pad injuries resulting from motorcycle wheel-spoke trauma, remains limited. This randomized controlled trial is designed to evaluate the efficacy of platelet-rich plasma dressing compared with saline dressing in children aged 5 to 12 years presenting with heel pad injuries.

A total of 60 participants will be enrolled and randomly assigned to receive either platelet-rich plasma dressing or saline dressing. Study outcomes will include wound healing within 12 weeks, duration of wound healing in days, and changes in wound size measured in both longitudinal and horizontal dimensions. This trial aims to generate evidence for a more effective and locally feasible wound management strategy for pediatric heel pad injuries in the study setting.

ELIGIBILITY:
Inclusion Criteria :

* Children aged 5-12 years
* Both genders
* Presenting with heel pad injuries caused by motorcycle wheel-spoke trauma

Exclusion Criteria :

* Children with wounds older than 3 weeks
* Children with wounds resulting from comorbidities

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Wound Healing Status | Up to 12 weeks
  Wound status based on presence of granulation tissue and measurement of wound size.

SECONDARY OUTCOMES:
Duration of healing | Up to 12 weeks
  Number of days from baseline until there is no further change in wound size.
Percentage Change in Longitudinal Wound Dimension | 12 weeks
  Calculated as (baseline longitudinal size - size at 12 weeks) ÷ baseline longitudinal size × 100.
Percentage Change in Horizontal Wound Dimension | 12 weeks
  Calculated as (baseline horizontal size-sizeat12weeks)÷base line horizontal size X 100

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected in this study will not be shared outside the study team to protect participant privacy and in accordance with local regulations.

REFERENCES:
- [Background] Somani A, Rai R. Comparison of Efficacy of Autologous Platelet-rich Fibrin versus Saline Dressing in Chronic Venous Leg Ulcers: A Randomised Controlled Trial. J Cutan Aesthet Surg. 2017 Jan-Mar;10(1):8-12. doi: 10.4103/JCAS.JCAS_137_16. PMID 28529414
- [Background] Elsaid A, El-Said M, Emile S, Youssef M, Khafagy W, Elshobaky A. Randomized Controlled Trial on Autologous Platelet-Rich Plasma Versus Saline Dressing in Treatment of Non-healing Diabetic Foot Ulcers. World J Surg. 2020 Apr;44(4):1294-1301. doi: 10.1007/s00268-019-05316-0. PMID 31811339